CLINICAL TRIAL: NCT05225506
Title: Support + High Intensity Functional Training for Parkinson's
Acronym: SHIFT-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Colleges of Health Education (Other)
Responsible Party: Principal Investigator, Reed Handlery, Assistant Professor, Arkansas Colleges of Health Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-2021-025
Record Dates: First submitted 2022-01-09; First posted 2022-02-04 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
Keywords: exercise; physical activity; parkinson
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Pre and post test with assessments at baseline and after 3 and 6 months of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): In this single group design, all participants will be provided with 6 months of twice weekly supervised group exercise.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise sessions will be one hour in duration and be a combination of resistance, aerobic, and balance exercise, with emphasis on movements specifically targeting common deficits seen in Parkinson's.

SUMMARY:
Parkinson's is the fastest growing neurological disorder in the world. With more people living with Parkinson's than ever before, there is an urgent need for interventions that improve health and reduce disability. High intensity exercise has shown to be superior to other forms of exercise in that it can slow symptom progression. High intensity exercise also reduces the risk of cardiovascular events. This is pertinent considering one in five people with Parkinson's will die from cardiovascular disease. While Parkinson's specific exercise programs across the U.S. continue to increase, there are still many communities with limited to no access, including Fort Smith, Arkansas. Here, there are no expert level centers within 100 miles and not a single community-based exercise program. This research will offer a community and group-based exercise program for participants with Parkinson's and their care partners.

DETAILED DESCRIPTION:
This study, Support + High Intensity Functional Training for Parkinson's (SHIFT-PD), will provide no-cost, twice weekly, group-based, adaptable exercise programming for people with Parkinson's and their care partners. All participants will be required to have physician or advanced practice provider clearance to exercise (please see attached medical release form). All participants will be evaluated by a physical therapist at no-cost prior to beginning the intervention to assess eligibility for the study (please see methodology section below). All eligible participants will complete a demographics questionnaire requesting participant age, sex, race/ethnicity, marital status, household income, primary means of locomotion, month and/or year of Parkinson's diagnosis (people with Parkinson's only), relationship to participant with Parkinson's (care partner only). Demographic data will be utilized to describe the study population participating in the research study and to evaluate barriers and facilitators for participation. All eligible participants will undergo a battery of baseline outcome assessments prior to undergoing the exercise intervention.

Participants will participate in a maximum of twice weekly group-based exercise classes for up to 6 months. All exercise programming will be led by licensed physical therapists at a local gym, CrossFit Fort Smith. All physical therapists will be CPR/BLS certified and an automated external defibrillator will be available onsite. Exercise classes will incorporate aerobic, resistance, and/or balance training. Exercise intensity will be monitored by participant vital signs and/or participant Rating of Perceived Exertion. SHIFT-PD will follow all state, federal, and CDC guidelines regarding COVID-19 precautions.

ELIGIBILITY:
Inclusion criteria for people with Parkinson's

* Participants must be at least 18 years of age
* Participants must have a diagnosis of Parkinson's disease
* Participants must be able to communicate and read in English
* Participants must have physician or advanced practice provider clearance to exercise
* Participants must provide their own transportation to and from the research study
* Participants must be able to ambulate independently and/or propel a power or manual wheelchair independently

Inclusion criteria for people who identify as care partners of those with Parkinson's

* Participants must be at least 18 years of age
* Participants must be able to communicate and read in English
* Participants must have physician or advanced practice provider clearance to exercise
* Participants must be a self-identified care partner of a person with Parkinson's participating in the study
* Participants must provide their own transportation to and from the research study
* Participants must be able to ambulate independently and/or propel a power or manual wheelchair independently

Exclusion Criteria:

-Failure to meet above listed inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Participant Attendance at 6 months | After 6 months of exercise intervention
  The percentage of interventions sessions attended by participants.

SECONDARY OUTCOMES:
Change in lower extremity functional strength at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  Lower extremity strength will be measured via functional test (Five Times Sit to Stand). This test records the amount of time taken to rise and sit to and from a chair five consecutive times. Faster times indicate greater lower extremity strength.
Change in grip strength at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  Grip strength will be measured via hand held dynamometry. Participants will perform three trials using their dominant hand. The force of each grip will be recorded and averaged in pounds.
Change in Activities Specific Balance Confidence (ABC) Scale at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  The ABC scale is a 16-item participant-reported measure of balance confidence while performing various activities. Participants rank their level of confidence from 0 (not at all confident) to 100 (completely confident); scores from each item are then averaged for one final score. The maximum score is 100%, indicating high balance confidence.
Change in Parkinson's Disease Questionnaire - 39 (PDQ-39) at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  The PDQ-39 is a 39-item participant-reported questionnaire which assesses health-related quality of life across 8 domains (mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, bodily discomfort). Participants respond to each item using a 5-point Likert scale from 0 (never) to 4 (always). Items in each domain are scored by expressing summed item scores as a percentage (ranging from 0 to 100%). Lower scores indicate better quality of life.
Change in Mini Balance Evaluation Systems Test (Mini BESTest) at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  The Mini BESTest is a 14-item test that assesses Anticipatory balance, reactive postural control, sensory orientation and dynamic gait. Performance for each item is ranked on a 3-point ordinal scale (0,1, or 2) with a total possible score of 28 (indicating good balance).
Change in fast-paced gait speed at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  Fast-paced walking speed will be measured via 10 meter walk test, which has individuals walk 10 meters with the middle 6 meters timed; three trial are performed and the average time is taken. Faster walking speeds indicate greater mobility with walking.
Change in casual gait speed at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  Walking speed will be measured via 10 meter walk test, which has individuals walk 10 meters with the middle 6 meters timed; three trial are performed and the average time is taken. Faster walking speeds indicate greater mobility with walking.
Change in Social Support for Exercise Scale at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  The Social Support for Exercise Scale contains 13 items and asks participants to rank frequency of supporting exercise behaviors amongst both family and friends on a 5-point Likert scale (1, none to 5, very often). Scores range from 13 to 65 with higher scores indicating greater social support for exercise.
Change in Self efficacy for exercise scale at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  The Self-Efficacy for Exercise Scale contains 9 items and asks participants to rank their confidence (0, not confident to 10, very confident) in their ability to exercise three times per week for 20 minutes in 9 different scenarios. Scores range from 0 to 90 with higher scores indicating greater exercise self-efficacy.
Change in 6 Minute Walk Test at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  The 6 Minute Walk Test measures a participants ability to cover as much distance (measured in meters) as possible while walking for 6 minutes. Participants will walk along a pre-defined pathway for 6 minutes, resting as needed. The test is a measure of walking endurance with further distances indicating greater endurance.
Change in Rand 36-Item Health Survey at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  Health related quality of life will be measured via Rand 36-item Health Survey. This 36 item survey asks participants about their health in several categories (physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain and general health). Scores in each category are averaged and range from 0 to 100, with higher scores indicating better health-related quality of life.
Change in Movement Disorder Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  The MDS-UPDRS measures disability as a result of Parkinson's and allows tracking for progression of the disease. The scale has four parts (1, mentation, behavior and mood, 2, activities of daily living, 3, motor examination, and 4, complications of therapy. Each parkinsonian sign or symptom is ranked on a 5-point Likert scale (ranging from 0 to 4) with higher scores indicating greater impairments. The minimum score on the entire scale is 0 and the maximum is 199.
Change in Global Rating of Change at 6 Months | After 6 months of exercise intervention (T3)
  Participants will rate their perceived level of change on a 15-point Likert Scale ranging from -7 (a very great deal less/worse to +7 (a very great deal more/better) with 0 representing no change. They will use this scale to answer 6 separate questions: 1) amount of physical activity performed in an average week, 2) ability to walk leisurely, 3) ability to walk fast, 4) ability to walk for a long period of time, 5) ability to stand up from a seated position, 6) ability to steady yourself and prevent a fall.
Change in Self-Reported Physical Activity Level at 6 Months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  Participants report their perceived physical activity levels compared to people their own age using a 5-point Likert Scale ranging from "much more active" to "much less active".
Change in accelerometer-measured moderate-to-vigorous physical activity at 6 months | Prior to exercise intervention (T1), after 3 months of intervention (T2), and after 6 months of exercise intervention (T3)
  Physical activity levels will be measured via thigh-worn accelerometer (activPAL). This small device will be worn on the less affected thigh (or right thigh for care partners) of participants with Parkinson's. The activPAL is able to detect acceleration and body position (i.e. sitting, standing, or lying). Through collecting acceleration data, different intensities of physical activity will be inferred (i.e light, moderate and vigorous intensity physical activity), with moderate-to-vigorous intensity physical activity being used as the primary outcome measure. At all time points, participants will wear the activPAL for 7 consecutive days. The activPAL will be waterproofed and will not need to be removed for activities such as bathing.
Participant Retention | After 6 months of exercise intervention (T3)
  The number and percentage of participants who remain in the study through the final measurement point at 6 months.
Participant Recruitment Rate | Throughout the 6-month study period
  The number of participants recruited will be reported as a percentage of total participants contacted for study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Reed Handlery, PhD, Principal Investigator — Arkansas Colleges of Health Education
Locations (1):
- Arkansas Colleges of Health Education, Fort Smith, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benka Wallen M, Franzen E, Nero H, Hagstromer M. Levels and Patterns of Physical Activity and Sedentary Behavior in Elderly People With Mild to Moderate Parkinson Disease. Phys Ther. 2015 Aug;95(8):1135-41. doi: 10.2522/ptj.20140374. Epub 2015 Feb 5. PMID 25655884
- [Background] Pennington S, Snell K, Lee M, Walker R. The cause of death in idiopathic Parkinson's disease. Parkinsonism Relat Disord. 2010 Aug;16(7):434-7. doi: 10.1016/j.parkreldis.2010.04.010. Epub 2010 May 31. PMID 20570207
- [Background] Schenkman M, Moore CG, Kohrt WM, Hall DA, Delitto A, Comella CL, Josbeno DA, Christiansen CL, Berman BD, Kluger BM, Melanson EL, Jain S, Robichaud JA, Poon C, Corcos DM. Effect of High-Intensity Treadmill Exercise on Motor Symptoms in Patients With De Novo Parkinson Disease: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):219-226. doi: 10.1001/jamaneurol.2017.3517. PMID 29228079
- [Background] Uc EY, Doerschug KC, Magnotta V, Dawson JD, Thomsen TR, Kline JN, Rizzo M, Newman SR, Mehta S, Grabowski TJ, Bruss J, Blanchette DR, Anderson SW, Voss MW, Kramer AF, Darling WG. Phase I/II randomized trial of aerobic exercise in Parkinson disease in a community setting. Neurology. 2014 Jul 29;83(5):413-25. doi: 10.1212/WNL.0000000000000644. Epub 2014 Jul 2. PMID 24991037
- [Background] Ellis T, Boudreau JK, DeAngelis TR, Brown LE, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Dibble LE. Barriers to exercise in people with Parkinson disease. Phys Ther. 2013 May;93(5):628-36. doi: 10.2522/ptj.20120279. Epub 2013 Jan 3. PMID 23288910
- [Background] Ellis TD, Cavanaugh JT, DeAngelis T, Hendron K, Thomas CA, Saint-Hilaire M, Pencina K, Latham NK. Comparative Effectiveness of mHealth-Supported Exercise Compared With Exercise Alone for People With Parkinson Disease: Randomized Controlled Pilot Study. Phys Ther. 2019 Feb 1;99(2):203-216. doi: 10.1093/ptj/pzy131. PMID 30715489